CLINICAL TRIAL: NCT00132210
Title: Pegylated Interferon Therapy for Acute Hepatitis C Infection in HIV-infected Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Jürgen K. Rockstroh, Bonn University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BN-102/02
Record Dates: First submitted 2005-08-17; First posted 2005-08-19 (Estimated); Last update posted 2010-10-21 (Estimated); Status verified 2009-11

CONDITIONS: Hepatitis C; HIV Infections
Keywords: acute hepatitis C; HIV; pegylated interferon
MeSH Terms: conditions — Hepatitis C; HIV Infections | interventions — peginterferon alfa-2a; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: pegylated interferon — Pegylated interferon alfa-2a or -2b in standard dosage Ribavirin in case of genotype 1 or 4 at 1000 or 1200 mg/d according to body weight ist recommended.
  Other Names: Pegasys; PegIntron; Copegus; Rebetol

SUMMARY:
The purpose of this study is to determine whether pegylated interferon therapy is effective to treat acute hepatitis C infection in HIV-coinfected individuals.

DETAILED DESCRIPTION:
Background:HIV-infected individuals are at higher risk of developing a chronic course of hepatitis C after infection. Moreover, chronic hepatitis C is less well treatable in HIV-Coinfected than in hepatitis C monoinfected patients. There is basic research and clinical data on hepatitis C mono-infection supporting high sustained response rates of hepatitis C when treatment is started in the acute phase of infection.

Aim of the study: To determine whether pegylated interferon therapy is effective to treat acute hepatitis C infection in HIV-coinfected individuals.

Methods: Prospective, open-label, historical controlled trial. Eligible subjects are treated over 24 weeks with a pegylated interferon at standard dose. Weight-adjusted ribavirin comedication is recommended for HCV-genotypes 1 and 4. Treatment will be withheld for 12 weeks in order to allow spontaneous resolution in subjects with clinical symptomatic hepatitis C infection.

ELIGIBILITY:
Inclusion Criteria:

* Documented acute hepatitis C infection with detectable HCV-RNA (PCR-assay) and elevated serum alanine transferase (ALT) levels. An acute infection is defined by fulfilling two of the following 3 criteria within the preceding four months:

  1. known or suspected exposure to HCV,
  2. documented seroconversion to positivity for antibodies against HCV,
  3. a serum alanine transferase (ALT) level of more than 350 U/l with a documented normal level during the year before infection.
* Documented HIV-infection
* CD4 cells > 300 /µl
* Ability to understand and sign a written consent form
* Women of child-bearing age: negative pregnancy test

Exclusion Criteria:

* Autoimmune hepatitis or other autoimmune disease
* Decompensated liver disease
* Decompensated renal disease, i.e. creatinine clearance < 50 ml/min, according to Cockcroft-Gault
* Acute or chronic hepatitis B infection
* Acute infection with hepatitis A or other hepatotropic viruses
* New AIDS defining event less than 1 month prior to enrolment
* Malignancy other than cutaneous kaposi sarcoma treated with systemic chemo-therapy
* History of severe psychiatric conditions, in particular severe depression
* History of seizures
* History of organ transplantation
* Thyroid disease not medically compensable
* Severe heart disease
* Severe retinopathy
* Known allergy to the study drug or one of the galenic compounds
* Hypersensitivity to interferon a
* Thrombocytes < 90 G/l, neutrophils < 1.5 G/l, hemoglobin must not be < 12g/dl (female) or < 13 g/dl (male)
* Treatment with corticosteroids less than 3 months prior to enrolment
* Alcohol abuse or use of other recreational drugs
* Older than 65 years of age, younger than 18 years of age
* Pregnancy, breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2002-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Negative hepatitis C ribonucleic acid (HCV-RNA) in peripheral serum | Week 24
Normal liver enzymes | Week 24

SECONDARY OUTCOMES:
Negative HCV-RNA | Week 12 and 48
Normal liver enzymes | Week 12 and 48

CONTACTS AND LOCATIONS:
Overall Officials: Jürgen K Rockstroh, MD, PhD, Study Director — Medical Department I, University Hospital, Bonn University, Germany; Martin Vogel, MD, Principal Investigator — Medical Department I, University Hospital, Bonn University
Locations (14):
- Germany (14):
  - Practice Hintsche, Berlin
  - Practice Bieniek, Berlin
  - Practice Dupke/Carganico/Baumgarten, Berlin
  - Practice Schranz, Berlin
  - Practice Freiwald/Rausch, Berlin
  - Practice Jessen, Berlin
  - Practice Kluschke, Berlin
  - Ärzteforum Seestraße, Berlin
  - Practice Center Kaiserdamm, Berlin
  - Medical Department I, University Hospital, Bonn University, Bonn
  - Practice St. Georg, Hamburg
  - Practice Fenske, Hamburg
  - Practice Linnig, Hamburg
  - Practice Trein, Stuttgart

REFERENCES:
- [Background] Vogel M, Bieniek B, Jessen H, Schewe CK, Hoffmann C, Baumgarten A, Kroidl A, Bogner JR, Spengler U, Rockstroh JK. Treatment of acute hepatitis C infection in HIV-infected patients: a retrospective analysis of eleven cases. J Viral Hepat. 2005 Mar;12(2):207-11. doi: 10.1111/j.1365-2893.2005.00580.x. PMID 15720537
- [Result] Vogel M, Nattermann J, Baumgarten A, Klausen G, Bieniek B, Schewe K, Jessen H, Boesecke C, Rausch M, Lutz T, Fenske S, Schranzo D, Kummerle T, Schuler C, Theisen A, Mayr C, Seidel T, Rockstroh JK. Pegylated interferon-alpha for the treatment of sexually transmitted acute hepatitis C in HIV-infected individuals. Antivir Ther. 2006;11(8):1097-101. PMID 17302380